CLINICAL TRIAL: NCT03554928
Title: Longitudinal Assessment of Functional Connectivity in Treatment Engaged Cocaine Users
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Colleen A Hanlon, PhD, Associate Professor, Medical University of South Carolina
Other Study IDs: 33406
Record Dates: First submitted 2018-04-12; First posted 2018-06-13 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cocaine Dependence; Substance Use Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cocaine Dependent: Individuals with cocaine dependence
  Interventions: Diagnostic Test: magnetic resonance imaging
- Not Cocaine Dependent: Individuals without cocaine dependence
  Interventions: Diagnostic Test: magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: magnetic resonance imaging — Participants will receive a 60 minute magnetic resonance imaging assessment

SUMMARY:
High-relapse rates to addiction are likely due to motivational (limbic) and cognitive (executive) factors. The purpose of this proposal is to determine the relationship between functional connectivity in executive control regions (namely the dorsolateral prefrontal cortex) and both proximal and extended outcomes in treatment seeking cocaine and opiate users. This longitudinal neuroimaging study will assess the integrity of executive and limbic circuits 4 timepoints before and after a 28-day intensive outpatient treatment program. Controls will also be recruited as a comparison group. The fundamental neuroscience knowledge gained from this proposal will be used to develop new evidence-based brain stimulation treatment strategies to enhance the integrity of these circuits and subsequent outcomes in traditional treatment programs.

The purpose of this study is not only to look at the integrity of these circuits in individuals entering treatment but also to see how these circuits change after treatment and if this can be used to predict outcomes. From the larger societal perspective this research may help us determine which individuals are likely going to benefit the most from treatment and perhaps those that are at a greater risk for relapse.

DETAILED DESCRIPTION:
Chronic cocaine use is among the most difficult substance-use disorders to treat. High relapse rates are likely due to a combination of factors that involve limbic and executive circuits in the brain, including vulnerability to salient cues and loss of cognitive control . This may be due to elevated functional activity within limbic neural circuitry, in the presence of a salient cue or to attenuated activity in executive control circuitry, which is impaired in users and is likely required to resist the limbic drive to use cocaine among individuals trying to remain abstinent.

Although predicting cocaine relapse after traditional outpatient treatment programs has largely focused on behavioral metrics, emerging literature suggests that neurofunctional activity may be a more robust predictor of relapse. While drug cue-reactivity in limbic processing regions (including the medial prefrontal cortex (MPFC), insula, and striatum) may predict relapse, activity in executive control regions (including the dorsolateral PFC (DLPFC)) is associated with sustained abstinence . Specifically, individuals that remain abstinent for 3 or more months have higher PFC gray matter integrity and baseline functional activity in their PFC relative to active users or recently abstinent peers . Most of these studies however are cross-sectional and assess these brain regions in isolation rather than as integrated networks.

Through interleaved transcranial magnetic stimulation (TMS) in the MRI environment, it is possible to differentially activate executive control and limbic circuitry by applying pulses of stimulation to the dorsolateral PFC (DLPFC) and MPFC respectively [31]. Extending decades of knowledge about the top-down influence of executive control circuitry on limbic circuitry, functional connectivity analysis revealed that TMS-induced DLPFC activity is negatively correlated with frontal and striatal elements of limbic circuit activity, including the medial and orbital PFC and the caudate. This 'negative' functional connectivity between the DLPFC and limbic regions however, was not present in a cohort of cocaine users with a history of relapse (see Significance). The overarching goal of this longitudinal imaging study is to use the novel probe to determine the relationship between executive and limbic circuit integrity as it relates to immediate and extended outcomes after an intensive outpatient treatment program. This will be achieved by assessing functional connectivity in treatment-seeking cocaine users and non-drug using controls at baseline (Aim1), and after a 28-day cognitive-behavioral treatment program (users only)(Aim 2). The relationship between the integrity of these circuits and clinically meaningful outcome measures will be determines 60 days and 90 days after baseline (Aim 3).

Aim 1: Investigate baseline executive and limbic circuit connectivity in treatment-seeking users and controls. Hypothesis: Interleaved imaging will demonstrate that cocaine users (n=55) have significantly lower % signal change in the DLPFC than controls, lower positive connectivity between the DLPFC (low integrity of executive circuitry) and the dorsal striatum, and lower negative connectivity between the DLPFC and the MPFC (low executive influence on limbic circuitry), suggesting that the DLPFC does not effectively modulate limbic circuitry in cocaine users.

Aim 2: Quantify changes in executive and limbic circuit connectivity that may occur following a 28-day cognitive-behavioral treatment program. Hypothesis: Cocaine users will have an elevation in the % signal change in the DLPFC (relative to Aim1), and the functional connectivity between the DLPFC and the limbic circuitry will increase (elevated influence of executive on limbic circuitry). Secondary hypothesis: This change in functional connectivity will be associated with a change in cognitive control on a battery of tests.

Aim 3: Determine the extent to which functional connectivity at baseline (Aim 1) or after treatment (Aim 2) is related to clinically-relevant metrics of drug use, cognitive control, and sustained connectivity after treatment commencement. Hypothesis: Within the 55 cocaine users, individuals that have the highest DLPFC % signal change or the highest negative correlation coefficient between the DLPFC and MPFC (at baseline and immediately after treatment), will be the individuals with the lowest number of drug positive urines, and will be the most likely to remain in the sample after 60 and 90 days of abstinence.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in an intensive outpatient treatment program for cocaine dependence

Exclusion Criteria:

* metal in the body below the neck
* history of traumatic brain injury

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals enrolled in an intensive outpatient rehabilitation program will be invited to enroll in this observational study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-06-09 (Actual); Study Completion 2019-06-09 (Actual)

PRIMARY OUTCOMES:
Percent change of Blood oxygen level dependent (BOLD) signal in executive compared to limbic brain regions | This will happen at the baseline MRI scan (Day 1), the 2nd MRI scan (1 month after Day 1), the 3rd MRI scan (2 months after Day 1), the 4th MRI scan (3 months after Day 1)
  Blood oxygen level dependent signal will be measured in several areas of the brain

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A Hanlon, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared on the NIH neuroimaging biorepository at the conclusion of data analysis
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: These data will be shared within 6 months of the final enrollment and data analysis.
Access Criteria: Access is open to the public